CLINICAL TRIAL: NCT00060359
Title: A Dose-Escalating Phase I Study With an Expanded Cohort to Assess the Feasibility of CT-2103 and Carboplatin (NSC #214240) in Patients With Previously Untreated Epithelial Ovarian, Primary Peritoneal, or Fallopian Tube Carcinoma
Brief Title: Polyglutamate Paclitaxel and Carboplatin in Treating Patients With Ovarian Epithelial, Peritoneal, or Fallopian Tube Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOG-9914; NCI-2012-02532 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000301642; GOG-9914 (Other: Gynecologic Oncology Group); GOG-9914 (Other: CTEP); U10CA027469 (NIH)
Record Dates: First submitted 2003-05-06; First posted 2003-05-07 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2015-05

CONDITIONS: Fallopian Tube Carcinoma; Malignant Ovarian Mixed Epithelial Tumor; Ovarian Brenner Tumor; Ovarian Clear Cell Cystadenocarcinoma; Ovarian Endometrioid Adenocarcinoma; Ovarian Mucinous Cystadenocarcinoma; Ovarian Serous Cystadenocarcinoma; Primary Peritoneal Carcinoma; Stage III Ovarian Cancer; Stage IV Ovarian Cancer; Undifferentiated Ovarian Carcinoma
MeSH Terms: conditions — Fallopian Tube Neoplasms; Brenner Tumor; Ovarian Neoplasms | interventions — Carboplatin; paclitaxel poliglumex

ARMS (1):
- Treatment (paclitaxel poliglumex, carboplatin) (Experimental): DOSE-ESCALATION PHASE: Patients receive CT-2103 IV over 10 minutes and carboplatin IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 8 courses in the absence of disease progression or unacceptable toxicity.
  Cohorts of 3-6 patients receive escalating doses of CT-2103 until the MTD is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity during the first course of treatment.
  FEASIBILITY PHASE: Once the MTD of CT-2103 is determined, an additional 20-40 patients receive treatment at that dose level combined with carboplatin as above.
  Interventions: Drug: Carboplatin; Drug: Paclitaxel Poliglumex; Other: Pharmacological Study

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplat; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Paclitaxel Poliglumex — Given IV
  Other Names: CT-2103; Paclitaxel Polyglutamate; Paclitaxel-Polyglutamate Polymer; PG-TXL; Poly-L-Glutamic acid-Paclitaxel Conjugate; Polyglutamic Acid Paclitaxel; Xyotax
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase I trial is studying the side effects and best dose of polyglutamate paclitaxel when given together with carboplatin in treating patients with ovarian epithelial, peritoneal, or fallopian tube cancer. Drugs used in chemotherapy such as polyglutamate paclitaxel and carboplatin use different ways to stop tumor cells from dividing so they stop growing or die. Polyglutamate paclitaxel may be able to deliver the drug directly to tumor cells while leaving normal cells undamaged. Combining polyglutamate paclitaxel with carboplatin may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose (MTD) of polyglutamate paclitaxel in combination with carboplatin in patients with chemotherapy-naïve ovarian epithelial, primary peritoneal, or fallopian tube carcinoma.

II. Determine the feasibility of this regimen at the MTD in an expanded cohort of patients.

III. Determine the response rate and progression-free survival of patients treated with this regimen in the expanded cohort.

IV. Determine the toxicity profile of this regimen in these patients. V. Determine the pharmacokinetics and pharmacodynamics of this drug combination in these patients.

OUTLINE: This is an open-label, multicenter, dose-escalation study of polyglutamate paclitaxel (CT-2103) followed by a feasibility, multicenter study.

DOSE-ESCALATION PHASE: Patients receive CT-2103 IV over 10 minutes and carboplatin IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 8 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of CT-2103 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity during the first course of treatment.

FEASIBILITY PHASE: Once the MTD of CT-2103 is determined, an additional 20-40 patients receive treatment at that dose level combined with carboplatin as above.

Patients are followed every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed ovarian epithelial, primary peritoneal, or fallopian tube carcinoma

  * Stage III or IV
  * Optimal (no greater than 1 cm) or suboptimal residual disease after initial surgery
* The following histologic epithelial cell types are eligible:

  * Serous adenocarcinoma
  * Mucinous adenocarcinoma
  * Clear cell adenocarcinoma
  * Transitional cell carcinoma
  * Adenocarcinoma not otherwise specified
  * Endometrioid adenocarcinoma
  * Undifferentiated carcinoma
  * Mixed epithelial carcinoma
  * Malignant Brenner tumor
* No epithelial tumors of low malignant potential (borderline tumors)
* Surgery performed within the past 12 weeks
* Performance status - GOG 0-2
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* No active bleeding
* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST and ALT no greater than 2.5 times ULN (5 times ULN if liver metastasis)
* Alkaline phosphatase no greater than 2.5 times ULN (5 times ULN if liver metastasis)
* No acute hepatitis
* PT and PTT normal
* Creatinine no greater than 1.5 times ULN
* Cardiac conduction abnormalities (e.g., bundle branch block or heart block) allowed provided cardiac status has been stable for the past 6 months
* No myocardial infarction within the past 6 months
* No unstable angina
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No neuropathy (sensory or motor) grade 2 or worse
* No other invasive malignancies within the past 5 years except nonmelanoma skin cancer or localized breast cancer
* No active infection requiring antibiotics
* No circumstances that would preclude study completion or follow-up
* More than 3 years since prior adjuvant chemotherapy for localized breast cancer (must be free of recurrent or metastatic disease)
* More than 3 years since prior radiotherapy for localized cancer of the breast, head and neck, or skin (must be free of recurrent or metastatic disease)
* No prior radiotherapy to any portion of the abdominal cavity or pelvis
* No prior treatment, other than debulking surgery, for this cancer
* No prior treatment for another cancer that would contraindicate this protocol therapy
* No concurrent amifostine or other protective reagents

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2003-04; Primary Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Feasibility, in terms of incidence of DLT, as assessed by CTC version 2.0 | 84 days (first 4 courses)
Maximum tolerated dose (MTD) as assessed by CTC version 2.0 | 21 days

SECONDARY OUTCOMES:
Incidence of cumulative toxicity | 168 days (8 courses)
Pharmacokinetics and pharmacodynamics of conjugated taxanes, unconjugated paclitaxel and carboplatin, as assessed by serum and urine measurements | 84 days (courses 1-4)
Progression-free survival | Up to 5 years
Response | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Mark Morgan, Principal Investigator — Gynecologic Oncology Group
Locations (1):
- Gynecologic Oncology Group, Philadelphia, Pennsylvania, United States